CLINICAL TRIAL: NCT07311356
Title: Evalutation of the Prognosis and Quality of Life of Patients Hospitalized for Early-onset Anorexia Nervosa
Brief Title: Prognosis of Early-onset Anorexia Nervosa
Acronym: AM2P
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250984; 2025-A01680-49 (Other: ANSM)
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Anorexia Nervosa
Keywords: early-onset anorexia nervosa; quality of life; prognosis
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohorte AM2P: Completion of quality of life questionnaire, clinic

SUMMARY:
The AM2P study aims to evaluate the long-term prognosis and quality of life of patients with early-onset anorexia nervosa, assessed 4 to 9 years after hospitalization. Prognosis will be determined using a composite outcome measure based on questionnaire responses and health indicators, including body mass index (BMI). In addition, the study will examine the patients' overall physical condition both at the time of assessment and during the interval between their last hospitalization and the present evaluation.

DETAILED DESCRIPTION:
This study includes all patients who were hospitalized at Robert Debré Hospital in Paris between 2016 and 2021 for early-onset anorexia nervosa. During follow-up interviews, participants will complete a standardized set of questionnaires assessing their mental and physical health (EDE-Q, PHQ-9, MSI-BPD, GAD-7, and SF-12). The primary outcome is the evaluation of the severity of the eating disorder, measured with the EDE-Q. Secondary outcomes will be derived from the additional questionnaires and will include body mass index (BMI), menstrual status, follow-up data, general well-being, impact of the eating disorder, hospital readmission, suicide attempts, depressive symptoms, borderline personality traits, anxiety, quality of life, educational attainment, occupational status, and treatments received. We hypothesize that approximately 50% of patients will achieve remission three years after hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* First full hospitalization in the eating disorders unit (EDU) at Robert Debré Hospital and diagnosis of AMP from 2016 to 2021
* No objection from the minor to the study
* Proficiency and understanding of the French language
* Access to digital technology (computer, smartphone, tablet, etc.)

Exclusion Criteria:

* Primary diagnosis of ARFID, other unspecified eating disorder

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients suffering from early_onset anorexia nervosa
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Score of Eating Disorder Examination Questionnaire (EDE SQ) scale | 6 months
  the percentage of subjective cure

SECONDARY OUTCOMES:
Identification of predictive factors at admission for the trajectory (remission/relapse) | 6 months
  The number of hospitalizations related to anorexia nerovsa

CONTACTS AND LOCATIONS:
Overall Officials: Coline STORDEUR, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Robert Debre - AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided